CLINICAL TRIAL: NCT00102986
Title: Sex Differences in Lopinavir/Ritonavir Pharmacokinetics Among HIV-1-Infected Men and Women
Brief Title: Differences in Blood Levels of Lopinavir/Ritonavir in HIV Infected Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5223; ACTG A5223; 10026 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infections
Keywords: Kaletra; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir

SUMMARY:
Men's and women's bodies may process anti-HIV drugs differently. The purpose of this study is to determine the differences in blood levels of soft gel capsules and tablets of lopinavir/ritonavir (LPV/r) in HIV infected men and women.

DETAILED DESCRIPTION:
It is estimated that 50% of people living with HIV/AIDS worldwide are women. HIV infected women face different psychosocial issues than men, and their bodies may react differently to HIV treatment. However, most of the data on the safety and efficacy of antiretrovirals (ARVs) used in the treatment of HIV infection are from studies conducted primarily in men. LPV/r in tablet form was approved by the FDA in October 2005. This study will determine the differences in pharmacokinetics (PK) in men and women taking a soft gel capsule and a tablet formulation of LPV/r.

No ARVs will be provided by this study. In Step 1, participants will receive soft gel capsules of LPV/r. All Step 1 participants will be asked to join Step 2 of the study upon completion of Step 1. In Step 2, participants will receive tablets of LPV/r. During the study, participants in both Step 1 and 2 will take a treatment regimen of LPV/r twice daily and one or more of the following: a nucleoside reverse transcriptase inhibitor (NRTI), tenofovir disoproxil fumarate, or enfuvirtide. Medical and medication history, blood collection, and clinical assessments will occur at study screening for both Steps 1 and 2. Participants in both steps will be asked to complete a medication diary from study entry to the day of the PK visit. The PK visit will occur within 30 days of study screening; blood collection for PK analysis will also occur at this visit.

ELIGIBILITY:
Note: Step 1 enrollment ended as of 06/28/06.

Inclusion Criteria

* HIV infected
* Have taken twice-daily LPV/r (soft gel formulation for Step 1 participants and tablet formulation for Step 2 participants) for at least 14 days immediately prior to step screening and are willing to continue taking LPV/r until the PK visit of that step
* Have taken LPV/r in combination with at least one of the following for at least 14 days immediately prior to study step screening: zidovudine, lamivudine, emtricitabine, stavudine, abacavir sulfate, didanosine, zalcitabine, tenofovir disoproxil fumarate, enfuvirtide, AND are willing to continue taking them until the PK visit of that step
* Body weight of more than 50 kg (110 lbs) for Step 1 participants only

Exclusion Criteria:

* Non-nucleoside reverse transcriptase inhibitor or dual protease inhibitor regimen within 30 days prior to study entry
* Require certain medications
* Current drug or alcohol abuse that, in the investigator's opinion, may interfere with the study
* Serious illness requiring systemic treatment or hospitalization within 30 days of study screening
* Acute AIDS-related opportunistic infection within 90 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2005-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Lopinavir (LPV) area under the concentration-time curve (AUC) for 0 to 12 hours

SECONDARY OUTCOMES:
LPV maximum concentration (Cmax), concentration at 12 hours (C12h), and apparent oral clearance (CL/F)
LPV AUC for 0 to 12 hours, Cmax, C12h, CL/F, and participant's race and ethnicity
LPV AUC for 0 to 12 hours, Cmax, C12h, CL/F, participant's age, weight, and body mass index (BMI), and coadministration of TDF
LPV AUC for 0 to 12 hours, Cmax, C12h, CL/F, and graded signs and symptoms
LPV AUC for 0 to 12 hours, Cmax, C12h, CL/F, and graded gastrointestinal signs and symptoms (defined as nausea, vomiting, diarrhea, abdominal pain, and bloating)
ritonavir (RTV) AUC for 0 to 12 hours, Cmax, C12h, and CL/F
LPV/r AUC for 0 to 12 hours, Cmax, C12h, CL/F for both the soft gel capsule and tablet formulations

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Currier, MD, MSc, Study Chair — Center for AIDS Research and Education, University of California, Los Angeles
Locations (29):
- United States (28):
  - University of Southern California CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Harbor-UCLA CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - The University of Miami AIDS Clinical Research Unit (ACRU) CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Cincinnati CRS, Cincinnati, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Umeh OC, Currier JS. Sex Differences in HIV: Natural History, Pharmacokinetics, and Drug Toxicity. Curr Infect Dis Rep. 2005 Jan;7(1):73-78. doi: 10.1007/s11908-005-0026-9. PMID 15610674